CLINICAL TRIAL: NCT07101952
Title: Influence of Suture Material Used for Cesarean Section Hysterotomy Closure on the Frequency of Scare Niche Formation
Brief Title: Suture Material and C-Section Scar Niches: A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Basma Sakr, Assistant Professor of Obstetrics & Gynecology, Faculty of Medicine, Benha University, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RC 2-11-2024
Record Dates: First submitted 2025-07-13; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vicryl group (Active Comparator): In these patients, the Cesarean section hysterotomy was closed using a double-layer technique involving unlocked continuous running sutures. The first layer incorporated the decidua, which was then overlapped by the second. The suture material used for this closure was conventional multifilament Vicryl.
  Interventions: Other: Multifilament vicryl suture material
- Barbed absorbable synthetic monofilament group (Active Comparator): In these patients, the Cesarean section hysterotomy was closed using a double-layer technique involving unlocked continuous running sutures. The first layer incorporated the decidua, which was then overlapped by the second. The suture material used for this closure was barbed suture; which is absorbable synthetic monofilament polydioxanone with bars.
  Interventions: Other: Braded Suture material

INTERVENTIONS:
Other: Braded Suture material — The Cesarean section hysterotomy was closed using a double-layer technique involving unlocked continuous running sutures. The first layer incorporated the decidua, which was then overlapped by the second. The suture material used for this closure was barbed suture; which is absorbable synthetic monofilament polydioxanone with bars.
  Other Names: Absorbable synthetic monofilament polydioxanone with bars
  Arms: Barbed absorbable synthetic monofilament group
Other: Multifilament vicryl suture material — The Cesarean section hysterotomy was closed using a double-layer technique involving unlocked continuous running sutures. The first layer incorporated the decidua, which was then overlapped by the second. The suture material used for this closure was barbed suture; which is absorbable synthetic monofilament polydioxanone with bars.
  Arms: Vicryl group

SUMMARY:
Defective healing of the uterine wound after a Cesarean section (CS) can lead to the formation of a CS niche (CSN). The specific technique used for closure and the type of suture material chosen are often overlooked factors that might contribute to the development of these niches. This study aimed to compare how frequently CSNs occur when the CS hysterotomy is closed using barbed suture material versus conventional vicryl suture material, with assessments primarily done via transvaginal ultrasound (TVS).

The methodology involved closing the CS hysterotomy with a double-layer technique using unlocked continuous running sutures, where the first layer included the decidua and was overlapped by the second. Researchers evaluated several aspects, including the duration and feasibility of the hysterotomy closure, the grade of postoperative pain, and the length of hospital stay. Transvaginal ultrasounds were conducted monthly for three months post-operatively to monitor for CSN development and to gather descriptive measurements of any niches found. The absence of a CSN was considered an indicator of surgical success.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for CS delivery either on emergency or elective bases for singleton fetus in cephalic presentation;
* Patients were free of exclusion criteria;
* Patients who signed the written consent to participate in the study and attend the postpartum follow-up for three months.

Exclusion Criteria:

* Patients who had multiple pregnancy;
* Patients who had fetus in abnormal lie or presentation;
* Patients who had previous repair of CSN;
* Patients with uncontrolled DM or hypertension;
* Patients who had maintained on immunosuppressive therapies, had autoimmune disorders;
* Patients who refused to sign the written consent were excluded from the study.

Ages: 22 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Surgical Success Rate in Relation to Suture Material | 3.5 Months
  The comparison of the overall surgical success rate, defined by the absence of a Cesarean section niche (CSN), between groups using different suture materials, alongside the quantitative differences in descriptive metrics of any formed CSNs.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha university, Banhā, El Qalyoubia, Egypt